CLINICAL TRIAL: NCT06458621
Title: Static Posturographic Analysis for Different Weight Categories in Adolescents
Brief Title: Weight Categories and Center of Pressure Sway
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Dina S. Noaman, demonstrator for pediatrics and its surgery, Delta University for Science and Technology
Other Study IDs: Weight categories
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Underweight group (A):: This group will be underweight group according to BMI- for age percentile growth chart ranged from BMI-for-age < 5th percentiles.
- Normal weight group (B):: This group will be with normal weight according to BMI- for age percentile growth chart which ranged from BMI-for-age 5th to 85th percentiles
- Overweight group (C):: This group will be an overweight group according to BMI- for age percentile growth chart which ranged from BMI-for-age 85th to 95th percentiles
- Obese group (D):: This group will be obese group according to BMI- for age percentile growth chart which ranged from BMI-for-age > 95th percentiles and <99th percentile

SUMMARY:
This study will be conducted to investigate the impact of different weight categories of adolescents on the center of pressure displacement throughout posturographic analysis test

DETAILED DESCRIPTION:
-Several studies have reported that obesity affects postural stability through center of pressure displacement in (adult, elderly and children). However, there are no studies illustrate the effect of variant weight categories (obese, overweight, normal weight, underweight) on static balance and postural stability by posturographic analysis in adolescent at age (16-18) years old.

I-Subjects:

200 adolescents from both sexes will be assigned to this study. They will be selected randomly from a secondary school student and first level university students. They will be selected according to the following criteria:

Inclusion criteria:

* Their age will be ranging from 16 to 18 years.
* The sample will be selected according to (BMI-for Age percentile) growth charts according to CDC (Centers for Disease Control and Prevention) (appendix-1) (NCHS, 2014)
* All participant will be free from any musculoskeletal deformities.
* All participant is free of peripheral neuropathic diseases.
* They have no visual or auditory or vestibular disorders.
* They will able to understand, follow and execute instructions included in the testing analysis procedures

They will be assigned into four group of equal numbers according to (BMI) body mass index for age percentile obese group (n=50), overweight group (n=50), underweight group (n=50) and normal group weight (n=50). They will be assigned as following:

Underweight group (A):

This group will be underweight group according to BMI- for age percentile growth chart ranged from BMI-for-age < 5th percentiles.

Normal weight group (B):

This group will be with normal weight according to BMI- for age percentile growth chart which ranged from BMI-for-age 5th to 85th percentiles

Overweight group (C):

This group will be an overweight group according to BMI- for age percentile growth chart which ranged from BMI-for-age 85th to 95th percentiles

Obese group (D):

This group will be obese group according to BMI- for age percentile growth chart which ranged from BMI-for-age > 95th percentiles and <99th percentile

II-Instrumentations:

A) For selecting subjects:

Use the CDC (Centers for Disease Control and Prevention) growth charts for children and teens aged 2 through 20 years. Comparing body measurements with the appropriate age- and sex-specific growth chart enables health care providers to monitor growth and identify potential health- or nutrition-related problems. (NCHS/CDC, 2014)

B) For evaluation:

1. Electronic body weight scale: for weight and Height measurements 2. Force platform: FREEMED platform and FREESTEP software (Sensor Medica, Inc., Via Umberto Agnelli 11, 00012 Guidonia Montecelio, Rome, Italy) were validated for both balance and gait analysis

III- Procedures:

For sample selection:

For subjects' selection use electronic body scale TCS-200-RT:

1. Weight

   A platform electronic scale was used to determine weight (TCS-200-RT). The participants will wear minimum clothes (removed jacket, shoes, and jewelry), stand stationary in the middle of the scale's platform without touching anything, and their body weight will be evenly distributed on both feet
   * A stadiometer (TCS-200-RT) with a vertical scale of 2 m and a sliding headpiece will be used to measure height to the closest 0.5 cm. The participants' heights will be measured without their shoes on. Participants will stand in the Frankfort horizontal plane The barefoot with eyes open. Initially they were instructed to stand relaxed with their feet separated at a comfortable width (about shoulder-width apart) and arms at sides in hanged position along the body and looking straight ahead and ankle-to-ankle angle 45° , and with the feet in a tandem position. The back of the head, heels, buttocks, and scapulae will be all against the vertical surface of the stadiometer.

   Plate form method of analysis:
   1. Testing procedures:

      -The experiments will be conducted in a quiet room, the force platform will be positioned in the middle. During the static standing trial each subject will permitted to speak occasionally with a partner sitting or standing in front of him or her about 2 meters away at any subject chosen by him or her, the collected data during the 80 sec of the trials will be analyzed for a-p direction (COP a-p) and m-l direction (COP m-l)

      -The test protocols usually include a Sensory Organization Test (SOT), During the test the subject is instructed to stand still and quietly with eyes open or closed depending on which of the six tests is being administered. The subject performs multiple trials per test .

      the testing protocol is consisted of six trials: in the 1st trial is bilateral eye opened (EO) for 20 sec; in the 2nd trail is bilateral eye closed (EC) for 20 sec; in 3rd trial is unilateral RT leg with EO for 10 sec; in 4th trail is unilateral RT leg EC for 10 sec, in the 5th trail is unilateral LT leg with EO for 10 sec and in the 6th trail is unilateral LT leg EC for 10 sec. The total test duration is 80 sec
   2. Testing parameters (outcomes):

      The following parameters will be tested
      1. Anteroposterior (AP) sway length rang of COP trajectory on (Y-Axis) (Delta Y).
      2. Mediolateral (ML) sway length rang of COP trajectory on (x-Axis) (Delta X).
      3. Average COP speed or velocity.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranging from 16 to 18 years.
* The sample will be selected according to (BMI-for Age percentile) growth charts according to CDC (Centers for Disease Control and Prevention)(NCHS, 2014)
* All participant will be free from any musculoskeletal deformities.
* All participant is free of peripheral neuropathic diseases.
* They have no visual or auditory or vestibular disorders.
* They will able to understand, follow and execute instructions included in the testing analysis procedures.

Exclusion Criteria:

* All adolescent associated with any musculoskeletal deformities.
* All adolescent associated with any foot deformity.
* All adolescent had a previous foot orthopedic procedure.
* All adolescent has visual or auditory or vestibular disorder.
* All adolescent has peripheral neuropathy.
* Adolescent with morbid obesity BMI >99th for age percentile

Ages: 16 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: They will be assigned into four group of equal numbers according to (BMI) body mass index for age percentile obese group (n=50), overweight group (n=50), underweight group (n=50) and normal group weight (n=50). They will be assigned as following:
  Normal weight group (B):
  This group will be with normal weight according to BMI- for age percentile growth chart which ranged from BMI-for-age 5th to 85th percentiles
  Overweight group (C):
  This group will be an overweight group according to BMI- for age percentile growth chart which ranged from BMI-for-age 85th to 95th percentiles
  Obese group (D):
  This group will be obese group according to BMI- for age percentile growth chart which ranged from BMI-for-age > 95th percentiles and <99th percentile
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Delta (Y)AP sway /mm | Through study completion an average of 5 months
  The anteroposterior COP sway length is the total distance traveled by COP in AP axis during the test time . The smaller the delta (y) , the better is the postural stability. It is an effective evaluation index in numerous populations and balance condition.
Delta (X)ML sway /mm | Through study completion an average of 5 months
  Mediolateral COP sway is the total distance traveled by COP in ML axis during the test time . The smaller the delta (x) , the better is the postural stability. It is an effective evaluation index in numerous populations and balance conditions.
Average COP speed /mm.s | Through study completion an average of 5 months
  is calculated by dividing the COP path length by testing time. In addition to the total COP average velocity, the average COP velocity components in the AP and ML directions can also be calculated. COP speed is an indicator of the efficiency of the postural control system. The average COP speed value is small, which is considered a good performance of posture control

CONTACTS AND LOCATIONS:
Overall Officials: Dina demonstrator for pediatrics and its surgery delta university, Bachelor, Principal Investigator — Delta University for Science and Technology
Locations (1):
- Delta university, Gamasa, Dakahlia Governorate, Egypt